CLINICAL TRIAL: NCT05218915
Title: Effect of Glucagon-like Peptide 1 Receptor Agonist in Combination with Insulin on Glycaemic Variability and Time-in-range in Diabetic Kidney Disease: a Randomised Controlled Trial
Brief Title: Basal Plus GLP1-ra on Glycemic Variability in CKD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Elaine Chow (Other)
Responsible Party: Sponsor-Investigator, Elaine Chow, Clinical Assistant Professor, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGLP-DKD
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus; Diabetic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Nephropathies | interventions — dulaglutide; insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- GLP1-ra plus basal insulin (BGLP) (Experimental): Dulaglutide and insulin degludec in combination with CGM
  Interventions: Drug: Dulaglutide; Drug: Insulin Degludec; Device: Continuous glucose monitor
- Basal bolus insulin (BB) (Active Comparator): Insulin aspart/lispro and insulin degludec in combination with CGM
  Interventions: Drug: Insulin Degludec; Device: Continuous glucose monitor

INTERVENTIONS:
Drug: Dulaglutide — Dulaglutide once weekly subcutaneous
  Arms: GLP1-ra plus basal insulin (BGLP)
Drug: Insulin Degludec — Insulin degludec once daily
Device: Continuous glucose monitor — Dexcom G6 CGM system

SUMMARY:
To compare GLP-1 RA plus basal insulin (BGLP) versus basal-bolus (BB) insulin regimens on glycemic variability (GV) and time in range (TIR) in diabetes patients CKD stage 3-4

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus diagnosed for at least 6 months
2. Male or female age ≥ 18 years old and ≤ 75 years old.
3. Body mass index between 18 and 40 kg/m2 inclusive
4. HbA1c ≥ 6.5% and ≤ 9.0% at screening
5. Women who are not pregnant, lactating or planning a pregnancy during their participation in the clinical study.
6. Patients with CKD stage 3 or 4 as defined by estimated glomerular filtration rate between 15-59 ml/min/m2 by the modified Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation at screening
7. Willingness, ability and commitment to comply with the testing, procedure and follow-up outlined in this protocol including (but not limited to) and use of pre-specified glucose monitoring devices.
8. In the opinion of the investigator, absence of any physical limitations, addictive diseases, or underlying medical conditions (including mental health) that may preclude the patient from being a suitable study candidate.
9. Written informed consent to participate in the study provided by the patient.
10. Willing and capable of use of a continuous glucose monitor as judged by the investigator

Exclusion Criteria:

1. Type 1 diabetes
2. Currently pregnant, as demonstrated by a positive pregnancy test at screening or planning pregnancy
3. Treatment with GLP-1 RA or insulin degludec in the past three months
4. Any active acute or chronic disease or condition that, in the opinion of the investigator, might interfere with the performance of this study.
5. Any active acute or chronic infectious disease that, in the opinion of the investigator, would pose an excessive risk to study staff.
6. Current use or recent exposure to any medication that in the opinion of the investigator could have an influence on the patient's ability to participate in this study or on the performance of the test device.
7. Extensive skin changes/diseases that preclude wearing the CGM on normal skin at the proposed application sites (e.g., extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis).
8. Have a known allergy to medical-grade adhesives
9. Known current or recent alcohol or drug abuse
10. Diabetic ketoacidosis, hyperosmolar hyperglycaemic state or myocardial infarction in the six months prior to screening
11. Patients on renal replacement therapy or likely require kidney transplant or dialysis during the study period
12. Currently participating in another investigational study protocol where the testing or results may interfere with study compliance, diagnostic results, or data collection.
13. An identified protected vulnerable patient (including but not limited to those in detention, or a prisoner).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Glycemic variability | 16 weeks
  % coefficient of variation on blinded CGM

SECONDARY OUTCOMES:
percent time in range | week 16 and 26
  percent time 3.9-10 mmol/l on CGM
percent time below range | week 16 and 26
  percent time below 3.9 mmol/l and below 3.0 mmol/l
percent time above range | week 16 and 26
  percent time above 10 mmol/l and 13.9 mmol/l
HbA1c | week 16 and 26
  HbA1c
Self reported hypoglycemia | 26 weeks
  level 1,2 and 3 hypoglycemia, biochemically confirmed
Self monitored glucose profiles | 26 weeks
  Fasting and postprandial
Body weight | week 16 and 26
  Body weight
Insulin doses | week 16 and 26
  Insulin doses
eGFR | week 16 and 26
  estimated glomerular filrate rate by CKD-EPI equation
uACR | week 16 and 26
  urine albumin creatinine ratio
Diabetes Treatment Satisfaction | week 16 and 26
  Chinese version of Diabetes Treatment Satisfaction Questionnaire, higher score better

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No